CLINICAL TRIAL: NCT05631132
Title: May Noninvasive Mechanical Ventilation (NIV) and/or Continuous Positive Airway Pressure (CPAP) Increase the Bronchoalveolar Lavage (BAL) Salvage in Patients With Pulmonary Diseases?
Acronym: PAP+BAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2203
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2022-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; Interstitial Lung Disease
Keywords: Bronchoalveolar Lavage; Noninvasive Mechanical Ventilation; Continuous Positive Airway Pressure; Bronchoscopy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BAL + NIV (Experimental): Qualification for a specific type of ventilation (NIV or CPAP) will be carried out in a randomized manner by a specially created online platform. The procedure will be performed subsequently in the same segment of the opposite lung. Once the test is finished, the volume of BAL fluid that has been recovered will be measured.
  Interventions: Procedure: BAL + PAP
- BAL + CPAP (Experimental): Qualification for a specific type of ventilation (NIV or CPAP) will be carried out in a randomized manner by a specially created online platform. The procedure will be performed subsequently in the same segment of the opposite lung. Once the test is finished, the volume of BAL fluid that has been recovered will be measured.
  Interventions: Procedure: BAL + PAP

INTERVENTIONS:
Procedure: BAL + PAP — May noninvasive mechanical ventilation (NIV) and/or continuous positive airway pressure (CPAP) increase the bronchoalveolar lavage (BAL) salvage in patients with pulmonary diseases?

SUMMARY:
The objective of our project is to find procedures and/or parameters to predict the diagnostic recovery (≥ 60% of the administered fluid volume) of bronchoalveolar lavage (BAL) fluid before bronchoscopy and to assess the impact of using non-invasive mechanical ventilation (NMV) or continuous positive airway pressure (CPAP) to achieve diagnostic recovery in patients with chronic obstructive pulmonary disease (COPD) and interstinal lungs disease for whom BAL performed during ordinary bronchoscopy turns out to be non-diagnostic.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosed stable COPD (Stages 1-3) - experimental group; Patients with interstitial lung disease - experimental group
2. Former and current smokers with normal lung function - potential control group 1;
3. Never-smokers with normal lung ventilation - potential control group 2.

Exclusion Criteria:

1. No written, informed consent to participate in the research project.
2. Severe respiratory failure (SaO2 < 90%)
3. The patient qualified for home oxygen treatment or home mechanical ventilation
4. Severe heart failure (NYHA class IV)
5. COPD mMRC IV
6. Myocardial infarction in the last two weeks or unstable angina
7. Severe, particularly ventricular arrhythmias
8. Platelet count < 20,000/ul
9. INR > 2 or APPT > 36 sec
10. Very severe obstruction: forced expiratory volume in 1 second (FEV1) < 30% of predicted.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-04 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
May noninvasive mechanical ventilation (NIV) and/or continuous positive airway pressure (CPAP) increase the bronchoalveolar lavage (BAL) salvage in patients with pulmonary diseases? | 3 years
  Comparison of fluid recovery with BAL with and without NIV connection

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmunology Department, Katowice, Poland

REFERENCES:
- [Derived] Danel A, Tobiczyk E, Warcholinski A, Trzaska-Sobczak M, Swinarew A, Brozek G, Trejnowska E, Batura-Gabryel H, Jedynak A, Scala R, Barczyk A, Cofta S, Skoczynski S. May noninvasive mechanical ventilation and/ or continuous positive airway pressure increase the bronchoalveolar lavage salvage in patients with pulmonary diseases? Randomized clinical trial - Study protocol. Adv Med Sci. 2023 Sep;68(2):482-490. doi: 10.1016/j.advms.2023.10.009. Epub 2023 Nov 7. PMID 37945441